CLINICAL TRIAL: NCT00610571
Title: Phase I Trial of Oral Topotecan Plus Temodar in the Treatment of Patients With Malignant Gliomas
Brief Title: Ph I Oral Topotecan and Temozolomide for Patients With Malignant Gliomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Katy Peters (Other)
Collaborators: GlaxoSmithKline (Industry); Schering-Plough (Industry)
Responsible Party: Sponsor-Investigator, Katy Peters, Assistant Professor, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00003970; 5487 (Other: Old Duke IRB number)
Record Dates: First submitted 2008-01-28; First posted 2008-02-08 (Estimated); Last update posted 2013-10-25 (Estimated); Status verified 2013-10

CONDITIONS: Glioblastoma; Gliosarcoma; Anaplastic Astrocytoma
Keywords: Temodar; Temozolomide; Topotecan; Hycamtin; Malignant Gliomas; Brain tumor; Anaplastic astrocytoma; AA; GBM; Glioblastoma Multiform; Gliosarcoma
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Astrocytoma; Glioma; Brain Neoplasms | interventions — Topotecan; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Oral Topotecan and Temodar (Experimental): Two separate strata to accrue independently. Stratum 1: Patients taking receiving Dilantin, Tegretol, Trileptal or Phenobarbital. Stratum 2: Patients on anti-convulsants other than Dilantin, Tegretol, Trileptal or Phenobarbital or patients not on any anti-convulsants
  Interventions: Drug: Oral Topotecan and Temodar

INTERVENTIONS:
Drug: Oral Topotecan and Temodar — Temozolomide is taken by mouth once day, every day for 5 consecutive days at dose of 200 mg/m2/day.
  Oral Topotecan will be taken daily for 5 consecutive days beginning 12-24 hrs after 1st dose of Temozolomide. Dose escalation of Oral Topotecan will be carried out in cohorts of 3 new subjects beginning w dose level 1 @ 0.75 mg/m2/dose.
  Other Names: Temodar - Temozolomide; Topotecan - Hycamtin

SUMMARY:
Objectives:

* To determine the maximum tolerated dose of oral topotecan when administered with Temodar to patients with malignant glioma
* To characterize any toxicity associated with the combination oral topotecan and Temodar.
* To observe patients for clinical antitumor response when treated with oral topotecan and Temodar.

DETAILED DESCRIPTION:
Subjects are patients with glioblastoma (GBM), anaplastic astrocytoma (AA) or grade 3 or greater WHO astrocytic, oligodendroglial or mixed glial tumors, which were initially diagnosed by histologic examination of biopsy/resection. Modified classical "3+3" phase I design used to determine maximum tolerated dose of topotecan in combination with Temodar.

ELIGIBILITY:
Inclusion Criteria:

* Histology: GBM, AA or grade 3 or greater WHO astrocytic, oligodendroglial or mixed glial tumors which were initially diagnosed by histologic exam of biopsy/resection
* Age: > or equal to 18 years
* Performance Status: Karnofsky Performance Status > or equal to 60% at study entry.
* Renal Function: Serum creatinine < 1.5 mg/dl or creatinine clearance > 60 ml/dL.
* Hematologic Status: The following baseline studies will be required before entry: total granulocyte count > or equal to 1000/microliter; platelet count > 100,000/microliter
* Hepatic Function: Serum SGOT & total bilirubin < or equal to 2.5 times ULN.
* Note: All lab parameters must have been obtained within 1 week of registration
* Consent: Signed informed consent, approved by IRB, will be obtained prior to initiating treatment
* Corticosteroids: For patients currently on corticosteroids, patients should be on stable dose for 1 week prior to study entry, if clinically possible.
* Prior Therapy: Interval of at least 2 weeks between prior surgical resection or prior radiotherapy (XRT) or 1 week from completion of chemotherapy and all toxicities are < or equal to grade 1 & enrollment on this protocol unless there is unequivocal evidence of progressive disease.
* Patients with Reproductive Potential: Patients must agree to practice effective birth control measures while on study and for 2 months after completing therapy

Exclusion Criteria:

* Pregnant or breast feeding women or women or men with reproductive potential not practicing adequate contraception. This therapy may be associated with potential toxicity to the fetus or child that exceeds minimum risks necessary to meet health needs of mother
* Active infection requiring intravenous antibiotics
* Prior failure with either topotecan or temozolomide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2004-04; Primary Completion 2009-09 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
maximum tolerated dose | 6 months

SECONDARY OUTCOMES:
Safety & efficacy | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Katherine B Peters, MD, PhD, Principal Investigator — Duke Health
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

REFERENCES:
- See also: The Preston Robert Tisch Brain Tumor Center at DUKE — http://www.cancer.duke.edu/btc/